CLINICAL TRIAL: NCT06348433
Title: Efficacy Evaluation and Mechanism Study of Ketogenic Diet on Autism Spectrum Disorder in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: QL000003
Record Dates: First submitted 2024-03-21; First posted 2024-04-04 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Ketogenic diet
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Diet, Ketogenic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketogenic diet group (Experimental): The subjects were treated with ketogenic diet. Ketogenic diet is a formula diet with high fat, low carbohydrate, proper amount of protein and other nutrients.ASD behavioral intervention measures are designed to help ASD patients improve their social communication skills, communication skills, behavior and other difficulties. Common intervention methods of ASD behavior include cognitive behavioral therapy, social skills training and so on.
  Interventions: Other: Ketogenic diet
- Ordinary diet group (No Intervention): ASD behavioral intervention measures are designed to help ASD patients improve their social communication skills, communication skills, behavior and other difficulties. Common intervention methods of ASD behavior include cognitive behavioral therapy, social skills training and so on.

INTERVENTIONS:
Other: Ketogenic diet — Ketogenic diet is a formula diet with high fat, low carbohydrate, proper amount of protein and other nutrients.
  Arms: Ketogenic diet group

SUMMARY:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder, which is characterized by social interaction and communication defects, rigid repetitive behaviors, and often accompanied by speech development retardation. According to the report released by the Morbidity and Mortality Weekly Report (MMWR) of the Centers for Disease Control and Prevention (CDC), according to the statistical data analysis in 2020, one out of every 36 8-year-old children (2.76%) was confirmed to have autism spectrum disorder (ASD). This ratio is higher than that published in December 2021, when the prevalence rate of 8-year-old children was 1/44 (2.3%) according to the statistics in 2018. Although ASD has a high incidence, there is still a lack of effective treatment measures for autism at present. Drug treatment can only partially alleviate some related symptoms, such as irritability and aggressiveness. Other interventions mainly focus on behavioral and educational interventions, which have limited help to patients. The high cost also leads to a huge burden on families and health care systems. Therefore, finding targeted treatment measures and treatment mechanisms for ASD as soon as possible has become an urgent problem for us to solve.Faced with limited treatment options, as many as a third of parents try various dietary pattern interventions to help their autistic children. In recent years, ketogenic diet, as a diet mode with extremely low carbohydrate, high fat, proper amount of protein and other nutrients, has attracted wide attention. In this mode, increased lipolysis puts the body in a ketosis state, thus ensuring energy supply.Although ketogenic diet (KD) has been proved to be effective in reducing the core symptoms in autistic patients and mouse models, the specific mechanism of KD in autism spectrum disorder (ASD) is still not completely clear.This study aims to evaluate the efficacy of ketogenic diet in improving core symptoms, sleep disorders and gastrointestinal symptoms of ASD children, explore the changes of excitation/inhibition (dorsolateral prefrontal cortex) in prefrontal cortex of ASD children before and after ketogenic diet intervention, and try to reveal the mechanism of ketogenic diet in treating ASD.

DETAILED DESCRIPTION:
1. Experimental design

   First of all, ASD children who come from the outpatient department of pediatric care, Qilu Hospital, Shandong University and have the willingness to join the group are evaluated, and the three routine auxiliary examinations are improved, such as liver and kidney function, blood lipid, myocardial enzyme, hematuria screening for genetic metabolic diseases, EEG and other ketogenic diet-related examinations. ASD children who meet the entry conditions sign informed consent and complete Gastrointestinal Symptom Rating Scale (GSRS score), Children's Sleep Habit Questionnaire (CSHQ) and Spectral Magnetic Resonance(MRS). Children in ketogenic diet group are randomly divided into ketogenic diet group or ordinary diet group by doctors Children in the ordinary diet group can still eat according to the previous diet structure and mode, and are followed up by doctors throughout the whole process.

   During this period, children in ketogenic diet group should regularly check blood glucose and ketone values, and measure their height and weight. The outpatient follow-up time is the 30th and 90th days of participating in this project.
2. The subjects were treated with ketogenic diet. Ketogenic diet is a formula diet with high fat, low carbohydrate, proper amount of protein and other nutrients. In 1921, Wilder, an American doctor, first put forward the concept of "ketogenic diet", which was used to treat epilepsy in children and achieved remarkable results. After 100 years' development, ketogenic diet has evolved into a variety of diet schemes, among which four are recognized by scholars at home and abroad, namely classic ketogenic diet (classic KD), medium chain triglyceride diet (MCT diet), improved Atkins diet (improved MAD) and low glycemic index therapy (LGIT).We chose the classic ketogenic diet as the treatment plan.Its keto food (fat) g/non-keto food (protein and carbohydrate) g ratio is 4: 1, fat accounts for about 90%, protein is about 7%, and carbohydrates are about 3%, limiting calorie intake. Professional nutritionists will refer to the height and weight percentile value table of children and adolescents aged 0-18 to evaluate the growth and development of children. If the growth and development are within the standard range or low, the recommended hot card is the actual weight * Recommended per kilogram The intake of hot cards should be high. If the growth and development are higher than the standard range, the recommended hot cards should be the standard weight corresponding to the actual height * Recommend the intake of hot cards per kilogram, and combine the amount of exercise of the child and whether to take hormone drugs, etc. An individualized diet plan for its growth and development, after determining the hot card, the nutritionist will carry out individualized meals according to the child's food allergies and other conditions.

ELIGIBILITY:
Inclusion Criteria:

* It meets the diagnostic criteria of ASD in the fifth edition of American Diagnostic Statistical Manual of Mental Disorders;
* Sign informed consent/agree to use ketogenic diet.

Exclusion Criteria:

* There are diseases related to fatty acid metabolism disorder and abnormal biological oxidation;
* Children who fail to maintain proper nutrition or fail to cooperate;;
* There are obvious intracranial lesions, organic brain diseases, abnormal liver function, abnormal kidney function and cardiovascular diseases;
* There are metal implants or metal foreign bodies in the body.

Ages: 18 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-03-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Autism Behavior Checklist（ABC） | At the beginning of ketogenesis and three months after ketogenesis
  There are 57 items in Autism Behavior Checklist（ABC）, including 5 dimensions: sensation, communication, physical movement, language and self-care. The highest score of the whole scale is 158 points, and the lowest score is 0 points. The higher the total score of the scale, the more serious the autistic behavioral symptoms are.
Childhood Autism Rating Scale(CARS) | At the beginning of ketogenesis and three months after ketogenesis
  The highest score on the Childhood Autism Rating Scale(CARS) scale is 60 points， and the lowest score is 0 points. The higher the total score of the scale, the more serious the autistic behavioral symptoms are.

SECONDARY OUTCOMES:
Gastrointestinal Symptom Scale（GSRS) | At the beginning of ketogenesis and three months after ketogenesis
  The total score of the Gastrointestinal Symptom Scale（GSRS) ranged from 0 to 78 points, and the higher the score, the more severe the gastrointestinal symptoms of the patient.
Children's Sleep Habits Questionnaire（CSHQ) | At the beginning of ketogenesis and three months after ketogenesis
  The Children's Sleep Habits Questionnaire（CSHQ) is used to assess Children's sleep behaviors and problems, with a minimum score of 22 and a maximum score of 110. The higher the score, the worse the child's sleep quality.

OTHER OUTCOMES:
MRS | At the beginning of ketogenesis and three months after ketogenesis,
  Magnetic resonance spectroscopy (MRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Yu Wang, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No